CLINICAL TRIAL: NCT01390792
Title: Special Drug Use Investigation for Relenza® (Zanamivir) (Prophylaxis)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112316
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed zanamivir: Subjects prescribed zanamivir during study period
  Interventions: Drug: Zanamivir hydrate

INTERVENTIONS:
Drug: Zanamivir hydrate

SUMMARY:
The purpose of this post-marketing surveillance study is to collect information on efficacy and safety for prophylactic administration of zanamivir in clinical practice in family or persons living with patients with influenza virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the study population criteria

Exclusion Criteria:

* Subjects with a history of hypersensitivity to the ingredients of zanamivir

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: <Zanamivir prophylactic administration group> Subjects meeting all of the following criteria and starting prophylactic administration of zanamivir
  * family or persons living with patients with influenza virus infection
  * subjects meeting any of the following criteria, elderly subjects ( 65 years old and over), subjects with chronic cardiac disease, with metabolic disease (diabetes, etc.) or with renal dysfunction
  * unvaccinated persons during the applicable seasons
  * subjects whose consent to write influenza diary was obtained
  <Non-zanamivir prophylactic administration group>
  - subjects meeting all of the above criteria and NOT starting prophylactic administration of zanamivir
Sampling Method: Probability Sample
Enrollment: 622 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events in subjects treated with zanamivir | 11 days
Occurrence of influenza virus infection | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Keizo Matsumoto, Hideyuki Okano, Naomi Hasegawa, Ichiro Ohwaki, Shogo Inoshiri. Study on Preventive Effects of Zanamivir (Relenza) for Influenza. Medicine and Drug Journal. 2010;46(11):121-132.